CLINICAL TRIAL: NCT01763216
Title: Improving Mood in Assisted Living Settings Using a Cognitive Training Intervention
Brief Title: Improving Mood in Assisted Living Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marianne Smith (Other)
Responsible Party: Sponsor-Investigator, Marianne Smith, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201208786
Record Dates: First submitted 2013-01-03; First posted 2013-01-08 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Depressive Symptoms; Clinical Depression
Keywords: depressive symptoms; clinical depression; visual processing speed; anxiety; pain; health-related quality of life
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Road Tour (Experimental): Road Tour was designed to improve the efficiency and accuracy of visual information processing and the ability to perform complex visual attention tasks. It focuses on improving the speed and accuracy with which users identify and locate visual information using a divided attention format. Over time, the difficulty and complexity of each task is systematically increased as users attain specified performance criteria. Difficulty is increased by reducing visual stimuli duration, adding visual distracters, increasing similarity between target and distracter stimuli, and presenting visual targets over a broader spatial expanse.
  Interventions: Other: Road Tour
- Boatload of Crosswords (Sham Comparator): Boatload of Crosswords offers the user a choice between three puzzle sizes, three levels of complexity, and varying font sizes. It also provides optional help features that the user may select, like filling in a letter or word to minimize frustration levels often associated with puzzle completion. Boatload of Crosswords was chosen for this study because it is computerized, it is very popular and easy to use, and many older adults enjoy doing crossword puzzles. Boatload of Crosswords, however, does not improve speed of processing because it does not focus on central discrimination and peripheral target location. Indeed, Boatload of Crosswords is not designed to train on any aspect of cognitive ability associated with visual speed of processing.
  Interventions: Other: Boatload of Crosswords

INTERVENTIONS:
Other: Road Tour — Training dosage includes 10 hours at baseline, four hours of booster training at month five, and four hours of booster training at month 11.
  Other Names: Road Tour at http://www.positscience.com
  Arms: Road Tour
Other: Boatload of Crosswords — Training dosage includes 10 hours at baseline, four hours of booster training at month five, and four hours of booster training at month 11.
  Other Names: Boatload of Crosswords at http://www./boatloadpuzzles.com
  Arms: Boatload of Crosswords

SUMMARY:
Late-life depression levels are escalating, and include 24% of all tenants of Assisted Living (AL) settings. A promising, novel intervention is a computerized visual speed of processing training program known as Road Tour. Road Tour has been show to reduce depressive symptom levels and the risk of onset of clinical depression in community dwelling older adults. The investigators hypothesize that similar benefits will accrue to residents in AL settings.

To evaluate this the investigators will use a two-arm, parallel, randomized controlled trial (RCT) comparing Road Tour training to attention control using computerized crossword puzzles among 370 adults 55 years old or older who reside in 15-30 AL settings that are partnering with the investigators.

The investigators hypothesize that Road Tour participants will have improved cognitive processing speed, lower levels of depressive symptoms, lower likelihood of the onset of clinical depression, less anxiety, lower levels of pain symptoms, and better health-related quality of life. These outcomes will be assessed at baseline, post-training, six months, and one year.

DETAILED DESCRIPTION:
Late-life depression is a large, escalating public health problem that often interacts with other health conditions and leads to spiraling disability that simultaneously threatens independence and health-related quality of life (HRQoL), and increases health care costs. Depression affects 24% of older adults in AL settings, but rates of recognition and treatment are low and underscore the need for alternative depression prevention and treatment methods in AL. A novel and promising intervention is a computerized cognitive training program known as Road Tour, which has shown serendipitous benefits for reducing depression symptoms and the onset of suspected clinical depression consistent with Beck's model of cognitive depression. As a self-directed, user-friendly "game", Road Tour overcomes common attitudinal and resource-related barriers that impede treatment in AL settings, and holds considerable promise for interrupting the potential downward spiral of depression-related disability for 1 million AL elders.

The purpose of this study is to evaluate the effect of Road Tour on processing speed, depressive symptoms and suspected clinical depression, and depression-related comorbidities among AL residents in Iowa. The investigators will use a two-arm, parallel, RCT comparing Road Tour training to attention control using computerized crossword puzzles among 370 adults 55 years old or older. The investigators will actively engage 15-30 AL settings and their associated facilities as study partners who implement the training at their sites and assist with the evaluation process. The investigators will help each AL setting develop AL-specific recruitment and enrollment protocols, educate AL staff about the study, and oversee computerized training by participating residents, as well as their family members and AL staff.

The investigators' three specific aims are to: (1) establish the effect of Road Tour on improving cognitive processing speed in AL; (2) evaluate the effect of Road Tour on reducing depressive symptoms and the risk of onset of suspected clinical depression in AL; and, (3) evaluate the effect of Road Tour on the depression-related health outcomes of anxiety, pain, and HRQoL in AL.

Participants will receive 10 hours of computerized training over 5-6 weeks, and 4 hours of booster training at months 5 and 11, for a total of 18 hours of training. Outcomes are changes in the Useful Field of View (UFOV) test for speed of processing (Aim 1), changes in the 12-item Centers for Epidemiologic Studies Depression scale (CESD-12) and the 9-item Patient Health Questionnaire (PHQ-9) for depressive symptoms and suspected clinical depression (Aim 2), and changes in the Short Form 36-item Health-Related Quality of Life (HRQoL) Questionnaire (SF-36) for HRQoL, the Brief Pain Inventory (BPI) for pain, and 7-item Generalized Anxiety Disorder questionnaire (GAD-7) for anxiety (Aim 3). Data will be collected using telephone interviews at baseline, post-training (6-8 weeks), and at 26-weeks and 52-weeks. Linear mixed effect models that adjust for the clustering within AL settings will be used with main effects specified for treatment group and time, as well as their two-way interaction. This study is the first step in evaluating depression-related outcomes of using Road Tour in AL settings.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or older
* reside in one of the participating AL settings or affiliated sites
* capable of providing informed consent

Exclusion Criteria:

* self-reported insufficient visual acuity (with glasses) to use a computer
* self-reported physical inability to use a computer mouse and keyboard
* non-English speaking

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Changes in the Patient Health Questionnaire (PHQ-9) | baseline, post-training, six months, one year
  The PHQ-9 items reflect the nine Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) diagnostic criteria for major depression and are rated from 0=not at all to 3=nearly every day for a total score range of 0-27. Established cut-points are: 0-4= minimal depression; 5-9=mild depression; 10-14=moderate depression; 15 or greater = severe depression. Scores of 10 or more indicate suspected clinically significant depression. The PHQ-9 facilitates direct assessment of two hallmarks of major depression (prominent dysphoria and anhedonia) and comparison to another body of late life depression research.
Changes in the Centers for Epidemiological Studies Depression (CESD) 12-item scale | baseline, post-training, six months, one year
  A shorter version of the original CESD-20 that has been a gold standard for screening for depression in epidemiological, field, and public survey studies, and has very high reliability and validity. Because the CESD-12 was used in the Iowa Healthy and Active Minds Study (IHAMS) and the Advanced Cognitive Training for Independent Vital Elderly (ACTIVE) study, direct comparison of depression outcomes among AL participants in this study and community-dwelling subjects in those studies can occur. CESD-12 is composed of short statements scored from 0=rarely or none of time (less than 1 day per week) to 3=all of the time (5-7 days per week) for a score range of 0-36. The cut-off score for suspected clinical depression on the CESD-12 is 9 or more points, which is equivalent to 16 or more points for the CESD-20.

SECONDARY OUTCOMES:
Changes in the Useful Field of View (UFOV) | baseline, post-training, six months, one year
  The UFOV is well-established, has high reliability and validity, and is the gold standard for measuring visual processing speed. UFOV includes three subtests-stimulus identification, divided attention, and selective attention-each automatically scored from 17-500 ms reflecting the shortest exposure time at which the participant could correctly perform each subtest 75% of the time, with a composite ms outcome score ranging from 51-1500 ms. Scores represent the shortest display duration with which the respondent performs accurately on 75% of the trials.
Changes in the Short Form 36 Item Health-Related Quality of Life (SF-36) Scale | baseline, and one year
  The SF-36 is the most widely used measure of health-related quality of life, and consists of 36 items that make up eight subscales. Its reliability and validity are well established in the US and elsewhere. Subscale scores range from 0 for worst health to 100 for best health.
Changes in the Short Form 12 Item Health-Related Quality of Life (SF-12) | post-training and six months
  The SF-12 is an abbreviated version of the SF-36 health-related quality of life measure, and consists of 12 items that make up eight subscales. Its reliability and validity are well established in the US and elsewhere. Subscale scores range from 0 for worst health to 100 for best health. It is used here at post-training and six months to minimize respondent fatigue.
Changes in the Brief Pain Invention (BPI) | baseline, post-training, six months, one year
  The Brief Pain Inventory (BPI) multi-item severity and interference scales have been adopted for telephone use. It consists of likert scaled and thermometer response options. We will examine mean changes in both scales over time, as well as declines in pain scores > 30%, which are considered clinically meaningful.
Changes in the Generalized Anxiety Disorder (GAD-7) Questionnaire | baseline, post-training, six months, one year
  The highly reliable and valid 7-item Generalized Anxiety Disorder (GAD-7) scale rates the DSM-IV criteria for GAD with a response set ranging from 0=not at all to 3=nearly every day. Cut-points for the GAD-7 are comparable to the PHQ-9, with 0-4= minimal anxiety; 5-9=mild anxiety; and 10 or more=clinically significant anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Smith, Ph.D., Principal Investigator — University of Iowa
Locations (32):
- United States (32):
  - Lakeview Village Retirement, Amana, Iowa
  - The Fountains Senior Community Living, Bettendorf, Iowa
  - Carlise Center for Assisted Living, Carlisle, Iowa
  - Western Home Communities, Cedar Falls, Iowa
  - Irving Point Affordable Assistant Living, Cedar Rapids, Iowa
  - Keystone Cedars, Cedar Rapids, Iowa
  - Meth-Wick Community, Cedar Rapids, Iowa
  - Prairie Hills at Cedar Rapids, Cedar Rapids, Iowa
  - Bickford of Clinton, Clinton, Iowa
  - Woodlands Creek Active Retirement Community, Clive, Iowa
  - Petersen Commons Assisted Living Community of Marycrest, Davenport, Iowa
  - Ridgecrest Village, Davenport, Iowa
  - Silvercrest Garner Active Retirement Community, Davenport, Iowa
  - Senior Star at Elmore Place, Davenport, Iowa
  - Wesley Acres, Des Moines, Iowa
  - Valley View Village, Des Moines, Iowa
  - The Kensington Assisted Living Community, Fort Madison, Iowa
  - Legacy Senior Living Community, Iowa City, Iowa
  - University of Iowa Colleges of Nursing and Public Health, Iowa City, Iowa
  - Emerson Point, Iowa City, Iowa
  - Melrose Meadows, Iowa City, Iowa
  - Oaknoll Retirement Residence, Iowa City, Iowa
  - Bishop Drumm--Martina Place, Johnston, Iowa
  - Summit Pointe, Marion, Iowa
  - The Villages at Marion, Marion, Iowa
  - Iowa Veteran's Home, Marshalltown, Iowa
  - Lutheran Living Senior Campus, Muscatine, Iowa
  - Manor Health Care Center, Sigourney, Iowa
  - Prairie Hills Assisted Living, Tipton, Iowa
  - Friendship Village Retirement Community, Waterloo, Iowa
  - Simpson Memorial Home, Inc., West Liberty, Iowa
  - Highland Ridge Senior Living Community, Williamsburg, Iowa

IPD SHARING:
Plan to Share IPD: No